CLINICAL TRIAL: NCT00724737
Title: Presurgical Planning With Motion Corrected fMRI Mapping of Motor Cortex in Patients With Cerebral Tumors
Brief Title: Presurgical Planning With Functional MRI (fMRI) Mapping of Motor Cortex in Patients With Cerebral Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Boklye Kim, Primary Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM 00050205; NIH
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fMRI of the brain, no surgery (Active Comparator): Healthy volunteers will undergo an fMRI (functional MRI of the brain).
  Interventions: Procedure: functional MRI (fMRI) of the brain
- fMRI of the brain, presurgical (Experimental): Patients scheduled to have brain surgery will undergo an fMRI (functional MRI of the brain).
  Interventions: Procedure: Presurgical MRI

INTERVENTIONS:
Procedure: Presurgical MRI — People who are scheduled to have brain surgery with undergo a fMRI of the brain before surgery. This is a "functional" scan, meaning that subjects will be asked to perform tasks (such as finger tapping or picture identification) during the MRI scan.
  Arms: fMRI of the brain, presurgical
Procedure: functional MRI (fMRI) of the brain — Healthy subjects will be undergo a brain fMRI of the brain. fMRI is a "functional" scan, meaning that subjects will be asked to perform tasks (such as finger tapping or picture identification) during the MRI scan.
  Arms: fMRI of the brain, no surgery

SUMMARY:
The purpose of this study is to determine if functional MRI is precise enough to provide information about the location of brain functions in patients who have brain tumors. This might allow physicians to use a non-invasive procedure to assist with brain mapping prior to surgery

DETAILED DESCRIPTION:
The purpose of this study is to determine if fMRI is precise enough to be used in preoperative decision making for patients who have brain tumors. Before a patient has brain surgery to have the tumor removed, functional mapping of the brain takes place either intra-operatively or post operatively after a subdural grid implant has been placed. Mapping helps the surgeon determine which areas of the brain are responsible for different important body functions. During this mapping procedure the surgeon determines if they can safely remove all or part of a brain tumor. The investigators are hoping to show that fMRI is just as accurate in mapping out different areas of the brain, without having to utilize an invasive form of brain mapping.

ELIGIBILITY:
Inclusion Criteria:

* All patients with brain tumors and healthy volunteers

Exclusion Criteria:

* If patients are pregnant.
* If patients suffer from a significant degree of claustrophobia.
* If patients are claustrophobic and requires general anesthesia to complete the diagnostic MRI.
* Contraindications for an MRI due to surgeries and/or implantation of pacemakers or pacemaker wires, open heart surgery for placement of an artificial heart valve, brain aneurysm surgery, middle ear implants, hearing aids, braces or extensive dental work, cataract surgery or lens implant, any implanted mechanical or electrical device, implanted neurological stimulators or artificial limbs or joints.
* Contraindications from an MRI due to foreign metallic objects in the body such as: bullets, BBs, pellets, surgical magnetic metal clips, joint or bone pins, metal plates, shrapnel or any one who has a history of working near metal who could have metal shavings in their eyes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Determining whether fMRI mapping is as effective as invasive presurgical mapping. | 2 weeks
  Subjects will be followed for the duration of their hospital stay with an expected average of 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Boklye Kim, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No